CLINICAL TRIAL: NCT04429646
Title: A Prospective, Multicenter, Randomized, Active Controlled, Clinical Trial of the LAMax LAA Closure System Compared to the Watchman® LAAC Device for Subjects With Non-valvular Atrial Fibrillation to Reduce the Risk of Ischemic Stroke
Brief Title: LAMax Vs. Watchman LAAC Device for Subjects With Non-valvular AF to Reduce the Risk of Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: The Third Medical Center, Chinese People's Liberation Army General Hospital (Unknown); The Second Affiliated Hospital of Chongqing Medical University (Other); Ganzhou Municipal Hospital (Unknown); First Affiliated Hospital of Guangxi Medical University (Other); The Second Hospital of Hebei Medical University (Other); The First Hospital of Jilin University (Other); LanZhou University (Other); Second Affiliated Hospital of Nanchang University (Other); The First Affiliated Hospital of Nanchang University (Other); The First Municipal hospital of Ningbo (Unknown); Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other); Tianjin Medical University General Hospital (Other); ShenZhen KYD Biomedical Technology Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Jian'an Wang,MD,PhD, President of the Second Affiliated Hospital, School of Medicine, Zhejiang University & Chief of Cardiology, Second Affiliated Hospital, School of Medicine, Zhejiang University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SAHZJU CT019
Record Dates: First submitted 2020-06-06; First posted 2020-06-12 (Actual); Last update posted 2022-05-06 (Actual); Status verified 2022-05

CONDITIONS: Non-valvular Atrial Fibrillation
Keywords: Atrial Fibrillation; Left Atrial Appendage Closure; Ischemic Stroke
MeSH Terms: conditions — Atrial Fibrillation; Ischemic Stroke

STUDY DESIGN:
Intervention Model Description: Allocation: Randomized Intervention Model: Parallel Assignment Primary Purpose: Prevention Endpoint Classification: Safety/Efficacy Study Masking: Open Label
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LAMax left atrial appendage occluder (Experimental): Intervention device, LAMax left atrial appendage closure system
  Interventions: Device: Percutaneous left atrial appendage closure-LAMax
- Watchman (control) (Active Comparator): Intervention device, Watchman® LAA Closure Device
  Interventions: Device: Percutaneous left atrial appendage closure-Watchman

INTERVENTIONS:
Device: Percutaneous left atrial appendage closure-LAMax — Interventional device, LAMax left atrial appendage closure system
  Arms: LAMax left atrial appendage occluder
Device: Percutaneous left atrial appendage closure-Watchman — Interventional device, Watchman® LAA Closure Device
  Arms: Watchman (control)

SUMMARY:
This is a prospective, multicenter, randomized, active controlled, clinical trial to evaluate the safety and effectiveness of the LAMax Left Atrial Appendage (LAA) Closure System.

DETAILED DESCRIPTION:
This is a prospective, multicenter, randomized, active controlled, clinical trial to evaluate the safety and effectiveness of the LAMax Left Atrial Appendage Closure (LAAC) System. Subjects with non-valvular Atrial Fibrillation will be randomized in a 1:1 ratio to the Experimental Treatment Arm (LAMax LAAC system) or the Control Arm (Watchman LAAC system, Boston Scientific Inc., USA). The trial is designed to demonstrate that safety and effectiveness of the LAMax device are non-inferior to the Watchman device.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years old with non-valvular atrial fibrillation (AF) and CHA2DS2-VASc ≥2
* There is one of the following: (1) Not suitable for long-term standard anticoagulation treatment; (2) On the basis of long-term standardized anticoagulant therapy with warfarin, stroke or embolism still occurred; (3) HAS-BLED ≥ 3.
* Provide written informed consent and agree to comply with required follow-ups.

Exclusion Criteria:

1. . Patients with other diseases other than AF who need long-term warfarin anticoagulation therapy;
2. . Those who need selective cardiac surgery;
3. . Heart failure NYHA grade IV;
4. . AF caused by rheumatic valvular disease, degenerative valvular disease, congenital valvular disease, severe mitral stenosis, aortic stenosis, or other valvular diseases;
5. . The early onset of AF and paroxysmal AF with definite causes, such as secondary to coronary artery bypass grafting (CABG), hyperthyroidism;
6. . Patients with symptomatic carotid artery disease (such as carotid stenosis > 50%);
7. . Patients with acute myocardial infarction, unstable angina, or recent myocardial infarction < 3 months;
8. . Stroke or TIA within 30 days;
9. . Bleeding disease, coagulation-related diseases, and active peptic ulcer;
10. . Active endocarditis, vegetations, or other infections causing bacteremia or sepsis;
11. . Conditions may lead to difficulty in testing or significantly shorten the life expectancy of patients (< 1 year);
12. . Pregnant, lactating or planned pregnancy during the trial;
13. . Patients who have not reached the end of other clinical trials of drug or device;
14. . Hematological abnormality (WBC < 3 × 109 / L, HB < 90g / L, or platelet count < 50 × 109 / L or > 700 × 109 / L));
15. . Renal insufficiency (creatinine > 3.0mg/dl or 265.2umoi / L), and / or advanced renal diseases requiring dialysis;
16. . Severe liver dysfunction (AST / ALT is 5 times higher than the upper limit of normal value, or total bilirubin is 2 times higher than the upper limit of normal value);
17. . The investigator believes that the patient is not suitable to participate in the clinical trial.
18. . Left atrial appendage has been removed, post heart transplantation, post atrial septal repair, or post occluder implantation;
19. . Radiofrequency ablation in 30 days before and after the implantation of LAA occluder;
20. . Cardioversion within 30 days after the implantation of LAA occluder;
21. . Post prosthetic heart valve replacement;
22. . Allergic to or contraindication to metal nickel alloy, aspirin, clopidogrel, contrast agent, heparin and other anticoagulants, etc;
23. . Patients who have placed other instruments in the cardiovascular cavity and are unable to place the LAA occluder;
24. . LVEF（left ventricular ejection fraction ）<35%；
25. . Clear thrombus is found in the heart before device implantation;
26. . TEE examination: refer to Watchman LAAC requirement to measure the orifice diameter of LAA, the maximum diameter is less than 17 mm, or more than 31 mm;
27. . Patent foramen ovale with high risk;
28. . mitral stenosis with a valve area ≤ 2 cm2;
29. . left atrial diameter > 65mm, or pericardial effusion more than a small amount, the depth of local effusion > 10 mm;
30. . Contraindications to X-ray, or not suitable for TEE examination.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 236 (Actual)
Dates: Start 2019-04-20 (Actual); Primary Completion 2020-11-11 (Actual); Study Completion 2021-06-10 (Actual)

PRIMARY OUTCOMES:
Successful sealing of the LAA | 12 months post-implantation
  A composite rate of successful sealing of the left atrial appendage (defined as residual flow ≤ 5 mm) at the 12-month visit documented by transesophageal echocardiogram (TEE).
Ischemic stroke, TIA, or Systemic embolism | 12 months post-implantation
  A composite rate of ischemic stroke, TIA or systemic embolism.

SECONDARY OUTCOMES:
All stroke, systemic embolism, or cardiovascular/unexplained death | 12 months post-implantation
  A composite rate of all stroke, systemic embolism, or cardiovascular/unexplained death.
Incidence of MACCE events | 12 months post-implantation
  A composite rate of MACCE, includes all-cause mortality, stroke, device embolism, cardiac tamponade.
Major Bleeding post-device implant | 12 months post-implantation
  Major bleeding rate at 12 months post-implant: defined as Type 3a or greater based on the Bleeding Academic Research Consortium (BARC) definition.
Success rate of device collapse and reposition during implantation procedure | 0 day
  It is one of the measures to describe device performance during implantation procedure.
Rate of cardiac temponade during implantation procedure | 0 day
  It is one of the measures to describe the performance of device and delivery system during implantation procedure.
Success rate of delivering an occlusion device to the LAA by the delivery system | 0 day
  It is one of the measures to describe the performance of delivery system during implantation procedure.
Success rate of withdrawing a delivery system after LAAC | 0 day
  It is one of the measures to describe the performance of delivery system.
Device performance post-implantation | 12 months post-implantation
  A composite rate of device migration, embolization, regurgitation, perivalvular leak post-implantation.
Device success rate | 0 day
  A composite rate to describe that the device can be successfully delivered in place and successfully implanted, and angiography shows that the implanted device is in the right position, no residual flow or residual flow is less than 5 mm, and the delivery system can be successfully withdrawn.
Perioperative clinical success rate | 7 days post-implantation
  A composite rate to describe that the device's function is normal, including that it was successfully implanted, the residual flow was less than 5mm, the implanted device had no effect on mitral valve movement and pulmonary vein blood flow, and there was no major adverse event (MAE) at the time of discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Jian-an Wang, MD, PhD, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University; Dongxing Ma, MD, Principal Investigator — The Third Medical Center, Chinese People's Liberation Army General Hospital
Locations (12):
- China (12):
  - The First Hospital of Lanzhou University, Lanzhou, Gansu
  - The Second Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Ganzhou Municipal Hospital, Ganzhou, Jiangxi
  - The Second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The First Hospital of Jilin University, Changchun, Jilin
  - The Second Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang
  - The First Municipal hospital of Ningbo, Ningbo, Zhejiang
  - The Third Medical Center, Chinese People's Liberation Army General Hospital, Beijing
  - The Second Affiliated Hospital of Chongqing Medical University, Chongqing
  - Shanghai Ninth People's Hospital, Shanghai JiaoTong University School of Medicine, Shanghai
  - General Hospital of Tianjin Medical University, Tianjin

REFERENCES:
- [Derived] Fan Y, Ma D, Wang C, Luo J, Ling Z, Li S, Peng X, Zhang Z, Chu H, Wang J; investigators in the present study. A Membrane Modification Technique for Left Atrial Appendage Occlusion: A Multicenter Randomized Controlled Trial. JACC Asia. 2025 Mar;5(3 Pt 1):374-387. doi: 10.1016/j.jacasi.2024.12.008. Epub 2025 Feb 18. PMID 40049930